CLINICAL TRIAL: NCT06160895
Title: Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TQ-A3334 Tablet After Multiple Doses in Healthy Adult Subjects
Brief Title: A Clinical Trial of TQ-A3334 Tablet After Multiple Administration in Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQ-A3334-I-04
Record Dates: First submitted 2023-11-30; First posted 2023-12-07 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- TQ-A3334 tablets (once a day) (Experimental): TQ-A3334 tablets, administered once a day.
  Interventions: Drug: TQ-A3334 tablets
- TQ-A3334 placebo tablets (once a day) (Placebo Comparator): TQ-A3334 placebo tablets, administered once a day.
  Interventions: Drug: TQ-A3334 placebo tablets
- TQ-A3334 tablets (every other day) (Experimental): TQ-A3334 tablets, administered once every other day.
  Interventions: Drug: TQ-A3334 tablets
- TQ-A3334 placebo tablets (every other day) (Placebo Comparator): TQ-A3334 placebo tablets, administered once every other day.
  Interventions: Drug: TQ-A3334 placebo tablets
- TQ-A3334 tablets (every three days) (Experimental): TQ-A3334 tablets, administered once every three days.
  Interventions: Drug: TQ-A3334 tablets
- TQ-A3334 placebo tablets (every three days) (Placebo Comparator): TQ-A3334 placebo tablets, administered once every three days.
  Interventions: Drug: TQ-A3334 placebo tablets

INTERVENTIONS:
Drug: TQ-A3334 tablets — TQ-A3334 tablet is a Toll like receptor 7 (TLR7) agonist.
  Arms: TQ-A3334 tablets (every other day); TQ-A3334 tablets (every three days); TQ-A3334 tablets (once a day)
Drug: TQ-A3334 placebo tablets — TQ-A3334 placebo tablet is a placebo that has no effect on TLR7.
  Arms: TQ-A3334 placebo tablets (every other day); TQ-A3334 placebo tablets (every three days); TQ-A3334 placebo tablets (once a day)

SUMMARY:
This study is a randomized, double-blind, placebo-controlled Phase I clinical study of TQ-A3334 tablets in adult healthy subjects, and the trial is planned to enroll 60 healthy subjects.

The primary objective is to evaluate the safety and tolerability of multiple dosing of TQ-A3334 tablets in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form before the study, and fully understand the study content, process and possible adverse events;
* Be able to complete the study according to the requirements of the protocol;
* Male and female subjects aged 18 to 55 years (inclusive);
* Male subjects weigh not less than 50 kg, female subjects weigh not less than 45 kg, Body Mass Index (BMI) in the range of 18 ~ 28 kg/m2 (inclusive);
* No clinically significant medical history of cardiac, hepatic, renal, gastrointestinal, neurological, respiratory, psychiatric abnormalities and metabolic abnormalities;
* Subjects (including partners) are willing to voluntarily take effective contraception within 2 weeks before screening to 6 months after the last dose of study drug.

Exclusion Criteria:

* Female subjects who are breastfeeding or plan to conceive or have a positive serum pregnancy results during the screening or study period;
* A pre-existing or current neuropsychiatric, respiratory, cardiovascular, gastrointestinal, hematologic-lymphatic, hepatic or renal insufficiency, endocrine, or musculoskeletal disease or other condition which, in the judgment of the Investigator, may have an effect on drug metabolism or safety;
* Eye diseases, including fundus lesions;
* History of clinically significant infections, including upper respiratory tract infections (URTI) and lower respiratory tract infections (LRTI), requiring antibiotic or antiviral medication within 14 days prior to screening or during screening;
* Acute illness or concomitant medication from the screening phase until study drug administration;
* History of dysphagia or any gastrointestinal disorder that interferes with drug absorption;
* Abnormal and clinically significant findings on vital signs, physical examination, laboratory tests, 12-lead electrocardiogram, abdominal ultrasound, and chest radiographs during the screening period;
* Positive for HBsAg in Hepatitis B, Hepatitis C, Syphilis, and Human Immunodeficiency Virus (HIV) antigen/antibody;
* Have taken any medication that can alter liver drug enzyme activity within 28 days prior to screening;
* Received immunoglobulin or blood product therapy within 30 days prior to screening;
* Have taken an investigational drug or participated in a clinical trial of any drug within 3 months prior to screening;
* Have taken Any prescription, over-the-counter, vitamin product, or herbal medication within 2 weeks prior to screening;
* Use of any systemic cytotoxic or systemic immunosuppressive drug within 6 months prior to screening or during the study period, or use of any localized cytotoxic or localized immunosuppressive drug within 30 days or 5 half-lives, whichever is longer, prior to screening or during the study period;
* Have undergone surgery within 4 weeks prior to screening or who plan to undergo surgery during the study period;
* Have lost blood or donated more than 400 mL of blood within 2 months prior to screening;
* Potential blood collection difficulties, history of needle and blood sickness;
* Having any clear history of drug or food allergy, especially to ingredients similar to those of the study drug;
* Those who smoked more than 5 cigarettes/day or used an equivalent amount of nicotine or nicotine-containing products within 3 months prior to screening, or who were unable to discontinue the use of any tobacco-based products during the trial;
* Those who have a history of chronic alcohol abuse or who have consumed more than 14 units of alcohol per week within 3 months prior to screening or who are unable to abstain from alcohol for the duration of the test or who have a positive breathalyzer test for alcohol;
* Those with a history of drug abuse or a positive urine drug screen;
* Those who can not avoid xanthine-rich beverages or foods or other factors that may affect drug absorption, distribution, metabolism, excretion, etc., from at least 1 day prior to study dosing until the end of the study;
* Subjects who, in the opinion of the investigator, have other factors that were unsuitable for participation in this trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) | From patient enrollment to withdrawal, estimated to be around 1 month.
  Incidence of adverse events (AE) evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Severity of adverse events (AE) | From patient enrollment to withdrawal, estimated to be around 1 month.
  Severity of adverse events (AE) evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Incidence of serious adverse events (SAE) | From patient enrollment to withdrawal, estimated to be around 1 month.
  Incidence of serious adverse events (SAE) evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Severity of serious adverse events (SAE) | From patient enrollment to withdrawal, estimated to be around 1 month.
  Severity of serious adverse events (SAE) evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Tolerability after drug administration | From patient enrollment to withdrawal, estimated to be around 1 month.
  Tolerability is evaluated by the number of participants with abnormal laboratory examinations, vital signs, physical examination, electrocardiogram.

SECONDARY OUTCOMES:
Peak Time (Tmax) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The time required to reach the highest concentration (peak drug concentration) on the human blood concentration curve after administration.
Peak concentration (Cmax) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The highest blood drug concentration achieved after administration.
Plasma concentration-area under time curve (AUC0-24) | From 60 minutes before administration on Day 1 to 24 hours after the last administration.
  The area under the plasma concentration-time curve from the beginning of the first administration to 24 hours.
Plasma concentration-area under time curve (AUC0-24) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The area under the plasma concentration-time curve from the beginning of the first administration to the last measurable concentration point.
Plasma concentration-area under time curve (AUC0-∞) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  Extrapolated from the first administration to the area under the plasma concentration-time curve to infinity.
Apparent volume of distribution (Vd/F) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The ratio of the drug dosage in the body to the blood drug concentration when the drug reaches dynamic equilibrium in the body.
Clearance (CL/F) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  Ratio of drug clearance rate to administration concentration.
Elimination half-life time (t1/2) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The time it takes to reduce the concentration of drugs in the blood by half
Time of maximum concentration under steady state (Tmax,ss) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  Time required to reach steady-state peak concentration after administration.
Maximum concentration under steady state (Cmax, ss) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The highest blood drug concentration that occurs after reaching steady state.
Minimum concentration under steady state (Cmin, ss) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The lowest blood drug concentration that occurs after reaching steady state.
Plasma concentration at steady state (Cav, SS) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The plasma concentration at which the rate of administration and rate of elimination are in equilibrium.
Plasma concentration area under steady-state time curve (AUCss) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The area under the plasma concentration-time curve of the steady state.
Accumulation Index (Rac) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The ratio of steady-state blood drug concentration to blood drug concentration after the first administration.
Degree of fluctuation (DF) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The ratio of the difference between the maximum steady-state blood drug concentration and the minimum steady-state blood drug concentration to the average steady-state blood drug concentration.
Interferon-α concentration (IFN-α) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The change of subjects' blood IFN-α concentration from baseline.
Interferon-stimulated gene concentration (ISG) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The change of subjects' blood ISG concentration from baseline.
Interferon-gamma concentration (IFN-γ) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The change of subjects' blood IFN-γ concentration from baseline.
Tumor Necrosis Factor-α concentration (TNF-α) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The change of subjects' blood TNF-α concentration from baseline.
Interleukin-6 concentration (IL-6) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The change of subjects' blood IL-6 concentration from baseline.
Interleukin-2 concentration (IL-2) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The change of subjects' blood IL-2 concentration from baseline.
Monocyte Chemotactic Protein 1 concentration (MCP-1) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The change of subjects' blood MCP-1 concentration from baseline.
Interferon-inducible protein-10 concentration (IP-10) | From 60 minutes before administration on Day 1 to 72 hours after the last administration.
  The change of subjects' blood IP-10 concentration from baseline.
QT/QT interval | From 30 minutes before administration on Day 1 to 48 hours after the last administration.
  Level of change in QT/QT interval to evaluate the drug cardiotoxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China